CLINICAL TRIAL: NCT01150643
Title: Identification of Biomarkers Predicting Responsiveness to Rituximab in Follicular Lymphoma
Brief Title: Biomarkers in Samples From Patients With Follicular Lymphoma Treated With Rituximab
Status: Completed | Type: Observational
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CDR0000675681; ECOG-E4402T1
Record Dates: First submitted 2010-06-24; First posted 2010-06-25 (Estimated); Last update posted 2017-05-17 (Actual); Status verified 2017-05

CONDITIONS: Lymphoma
Keywords: stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Follicular | interventions — Gene Expression Profiling; Microarray Analysis; Polymerase Chain Reaction; Amplified Fragment Length Polymorphism Analysis; Immunohistochemistry

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective

INTERVENTIONS:
Genetic: gene expression analysis
Genetic: microarray analysis
Genetic: polymerase chain reaction
Genetic: polymorphism analysis
Other: immunohistochemistry staining method
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying the effects of rituximab in blood and tumor tissue samples from patients with cancer in the laboratory may help doctors learn more about the effects of rituximab on cancer cells. It may also help doctors identify biomarkers related to cancer.

PURPOSE: This research study is studying biomarkers in samples from patients with follicular lymphoma treated with rituximab.

DETAILED DESCRIPTION:
OBJECTIVES:

* Correlate immunoglobulin Fc receptor (FcγR) polymorphisms with response, response duration, and time to resistance in samples from patients with follicular lymphoma (FL) treated with single-agent rituximab on ECOG-E4402.
* Identify gene expression profiles that correlate with response, response duration, and time to rituximab resistance in these patients.
* Determine whether the FL microenvironment is predictive of initial response and duration of response to rituximab.

OUTLINE: DNA and RNA from banked peripheral blood mononuclear cells (PBMCs) and formalin-fixed paraffin-embedded (FFPE) tumor samples are analyzed for immunoglobulin-receptor polymorphism, gene expression profile, and follicular lymphoma microenvironment by real-time PCR, microarray hybridization, and IHC.

PROJECTED ACCRUAL: A total of 259 PBMC samples and 300 FFPE blocks will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosed with follicular lymphoma
* Treated on ECOG-E4402 comprising 1 of 2 different rituximab-dose strategies
* Banked peripheral blood mononuclear cells (PBMCs) and formalin-fixed paraffin-embedded (FFPE) tumor samples available

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Samples from patients enrolled on E4402 from whom samples were submitted for research
Sampling Method: Non-Probability Sample
Enrollment: 559 (Actual)
Dates: Start 2010-12-06 (Actual); Primary Completion 2011-01-06 (Actual); Study Completion 2011-01-06 (Actual)

PRIMARY OUTCOMES:
Correlation between FcγR polymorphisms and rituximab response, response duration, and time to resistance | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Brad S. Kahl, MD, Principal Investigator — University of Wisconsin, Madison